CLINICAL TRIAL: NCT00313976
Title: A Scandinavian, Randomized, Rater-blinded Study of Single and Double-dose Betaferon in Patients With Early Secondary Progressive Multiple Sclerosis
Brief Title: Study to Compare Double-dose Betaferon to the Approved Dose, for Patients With Early Secondary Progressive Multiple Sclerosis (SPMS)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91449; EudraCT: 2005-001540-23; 309560
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2008-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Early secondary progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Interferon beta-1b

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046)
- Arm 2 (Experimental)
  Interventions: Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046) — 250 micrograms every other day, subcutaneously for 104 weeks
  Arms: Arm 1
Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046) — 2x250 micrograms every other day, subcutaneously for 104 weeks
  Arms: Arm 2

SUMMARY:
The purpose of the study is to evaluate if the higher dose can give greater efficacy without negative impact on the adverse event profile for patients with early secondary progressive Multiple Sclerosis (SPMS).

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS for no less than one year and no longer than ten years
* Disease in the secondary progressive (SP) phase
* At least one relapse the last 3 years
* Treatment with an interferon for at least 6 months and with Betaferon for at least 3 months

Exclusion Criteria:

* Serious or acute heart disease
* Severe depression
* Serious or acute liver, kidney or bone marrow dysfunction
* Epilepsy not adequately treated
* Pregnancy or lactation
* Alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI): T2-lesions | At week 104

SECONDARY OUTCOMES:
Further Magnetic Resonance Imaging (MRI) parameters | At week 104
Relapses | At week 104
Changes in Expanded Disability Status Score (EDSS) and Multiple Sclerosis Impact Scale (MSIS) | At week 104
Hospitalizations | At week 104
Neutralizing antibodies | At week 104
Adverse events | At week 104

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Denmark (4):
  - Ask Contact
  - Copenhagen
  - Hillerød
  - Holstebro
- Stockholm, Sweden